CLINICAL TRIAL: NCT00441168
Title: A Phase 2, Multicentre, Randomised, Open-Label, Parallel Group Study to Evaluate the Safety and Efficacy of Velcade When Added to Adriamycin-Dexamethasone Treatment Versus Vincristine-Adriamycin-Dexamethasone Standard Treatment in Subjects With Multiple Myeloma Who Are Refractory to or Have Relapsed After Primary Therapy for Multiple Myeloma
Brief Title: Velcade (Bortezomib), Adriamycin Dexamethasone (PAD) or Vincristine Adriamycin Dexamethasone in Second Line Treatment of Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: TRIAL STOPPED due to a change in standard of care and the required patient numbers could no longer be achieved
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR011065; 26866138MMY2038 (Other: Janssen-Cilag International NV); 2006-001709-27 (EudraCT Number)
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; bortezomib; Cancer; Hematology; bone marrow; immunoglobulin; relapse; refractory; plasma cell; Velcade; adriamycin; dexamethasone; vincristine
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Recurrence | interventions — Doxorubicin; Bortezomib; Dexamethasone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAD Treatment (Active Comparator): vincristine in combination with adriamycin and dexamethasone
  Interventions: Drug: adriamycin; Drug: dexamethasone; Drug: vincristine
- PAD Treatment (Experimental): bortezomib in combination with adriamycin and dexamethasone
  Interventions: Drug: adriamycin; Drug: bortezomib; Drug: dexamethasone

INTERVENTIONS:
Drug: adriamycin — adriamycin: 9mg/m² intravenous (IV) push on days 1 to 4
Drug: bortezomib — bortezomib: 1.3 mg/m² intravenous (IV) bolus on days 1, 4, 8, and 11
  Arms: PAD Treatment
Drug: dexamethasone — dexamethasone: 40 mg daily days 1- 4/9-12/17-20 - cycle 1 / days 1-4/17-20 - subsequent cycle
Drug: vincristine — vincristine: 0.4mg IV push on days 1 to 4
  Arms: VAD Treatment

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of replacing vincristine with a drug called bortezomib (also known as "Velcade"or PS341) in the standard therapy vincristine, doxorubicin (not limited to, but formerly referred to under the tradename Adriamycin) and dexamethasone (VAD) in patients with multiple myeloma. Multiple Myeloma is the second most common cancer of the blood. Bortezomib is the first approved cancer treatment in a new class of medicines called proteasome inhibitors. It disrupts the cell cycle of the cell, affecting numerous biologic pathways, including those related to growth and survival of cancer cells. The treatment will be used as second line treatment, which means either the disease has returned after a period of improvement (relapse) or the disease did not respond to the initial treatment (refractory). Patients will receive either bortezomib (PS341), doxorubicin (Adriamycin) and dexamethasone (PAD) or the VAD standard therapy.

DETAILED DESCRIPTION:
Bortezomib, has been approved for use in patients with multiple myeloma, who have already received at least one prior treatment and whose disease is worsening on their last treatment and who have already undergone or are unsuitable for bone marrow transplantation. Bortezomib has significant activity in patients with relapsed multiple myeloma, its efficacy is increased with the addition of dexamethasone and it demonstrates synergy with doxorubicin. The VAD combination has been widely used in multiple myeloma and has demonstrated to be effective in relapsed patients. Based on previous trial results, it is hoped that bortezomib, in replacing vincristine in the VAD standard therapy, can improve the response to treatment of patients with multiple myeloma, with manageable side effects. This is an international, multicentre, randomised, open-label, parallel group study. About 212 patients will take part in the study. Patients will be treated with either bortezomib (PS-341), Adriamycin and Dexamethasone (PAD) or Vincristine, Adriamycin and Dexamethasone (VAD). There will be an initial 14 day screening period to evaluate if the patient is suitable for the study. After screening, eligible patients will be randomised to receive either PAD or VAD. Patients will receive therapy for up to 8 treatment cycles of 28 days each. After the treatment period, there will be a long-term follow-up period with monthly visits until disease progression or relapse. Thereafter follow-up will be continued by at least a phone call every other month. This long-term follow-up period will be performed for all patients until the last patient was treated and followed up for 1 year. Response to treatment will be assessed according to the European group for blood and marrow transplant criteria (EBMT). Disease burden will be monitored by measuring M-protein concentration in serum and in urine every 4 weeks until disease progression or relapse. Thereafter follow-up for survival will be continued every other month by at least a phone call. Safety will be assessed by monitoring of adverse events (AEs), vital signs, physical examination and clinical laboratory tests. Treatment with PAD or VAD will be for up to 8 cycles of 28 days each. Treatment beyond 6 cycles will be discussed on individual basis. Proposed dosages are: bortezomib 1.3 mg/m² intravenous (IV) bolus on Days 1, 4, 8, and 11; vincristine 0.4mg IV push on Days 1 to 4; doxorubicin 9mg/m² IV push on Days 1 to 4; dexamethasone in 1st cycle 40 mg daily on Days 1 to 4, 9 to 12 and 17 to 20, orally (or equivalent parenteral dose) and on subsequent cycles as 40 mg daily on Days 1 to 4 and 17 to 20 only.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma following 1 previous line of therapy and, is scheduled by the investigator to be treated with vincristine, adriamycin and dexamethasone standard therapy
* measurable secretory multiple myeloma based on defined criteria
* Karnofsky performance status of >or = 60%
* fulfils defined laboratory requirements within 14 days before baseline
* if female, the patient is either postmenopausal or surgically sterilised or willing to use an acceptable method of birth control for defined period of time
* if male, the patient agrees to use an acceptable barrier method for contraception for a defined period of time.

Exclusion Criteria:

* More than one previous line of therapy for multiple myeloma
* use of bortezomib in the previous line of therapy and/or received bortezomib in a previous trial
* known allergy or hypersensitivity to bortezomib, boron or mannitol
* peripheral neuropathy or neuropathic pain of grade 2 or higher
* myocardial infarction within 6 months of enrollment or had New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (16):
- Zagreb, Croatia
- Germany (2):
  - Leer
  - Velbert
- Debrecen, Hungary
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (3):
  - Bialystok
  - Gdansk
  - Poznan
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Samara
- Turkey (Türkiye) (3):
  - Ankara
  - Bursa
  - Eskişehir

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 05 December 2006 to 04 July 2007 at 2 sites in Germany, 1 site in Hungary, 3 sites in Lithuania, 3 sites in Poland and 3 sites in Russia
Pre-assignment Details: Subjects who qualified were screened. Subjects were considered for eligibility when the investigator would treat the subject with a combination therapy of vincristine, adriamycin and dexamethasone (VAD) standard therapy. One subject was not randomised because the subject was a screening failure.
Groups:
- VAD Treatment: vincristine: 0.4mg IV push on days 1 to 4; adriamycin: 9mg/m² IV push on days 1 to 4; dexamethasone: 40 mg daily days 1- 4/9-12/17-20 - cycle 1 / days 1-4/17-20 - subsequent cycle
- PAD Treatment: bortezomib: 1.3 mg/m² intravenous (IV) bolus on days 1, 4, 8, and 11; adriamycin: 9mg/m² IV push on days 1 to 4; dexamethasone: 40 mg daily days 1- 4/9-12/17-20 - cycle 1 / days 1-4/17-20 - subsequent cycle
Period: Treatment Period
Arm/Group | VAD Treatment | PAD Treatment
Started | 17 | 13
TREATED | 16 | 13
Completed | 6 | 7
Not Completed | 11 | 6
Not completed — Death | 3 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Progressive Disease | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — qualified for stem-cell transplantation | 3 | 0
Not completed — refractory disease | 1 | 0
Period: Follow-up Period
Arm/Group | VAD Treatment | PAD Treatment
Started | 17 (Subjects who did not complete the treatment period could be entered into the follow-up period) | 13 (Subjects who did not complete the treatment period could be entered into the follow-up period)
Completed | 5 | 4
Not Completed | 12 | 9
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAD Treatment | PAD Treatment | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.4) | 61.5 (11.3) | 62.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Karnofsky Performance Status [Number; unit: participants] — A standard way of measuring the ability of cancer patients to perform ordinary tasks. The Karnofsky Performance Scores (KPS) range from 0 to 100. A higher score means the patient is better able to carry out daily activities. KPS may be used to determine a patient's prognosis, to measure changes in a patient's ability to function, or to decide if a patient could be included in a clinical trial.
  participants
    ≤50 | 0 | 0 | 0
    60 | 1 | 1 | 2
    70 | 1 | 3 | 4
    80 | 9 | 3 | 12
    90 | 5 | 3 | 8
    100 | 0 | 3 | 3
Body Surface Area [Mean (Standard Deviation); unit: m2] | 1.855 (0.233) | 1.924 (0.219) | 1.886 (0.226)
Height [Mean (Standard Deviation); unit: cm] | 168.8 (11.2) | 169.8 (9.5) | 169.3 (10.3)
Weight [Mean (Standard Deviation); unit: kg] | 75.9 (15.7) | 78.3 (14.5) | 77.0 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Best Confirmed Disease Response
Description: The primary efficacy analysis was based on the best response obtained during the treatment period according to the European Group for Blood and Marrow Transplantation (EBMT) criteria as assessed by the investigator. The best confirmed response was defined as 2 separate and consecutive evaluations of response, at least 6 weeks apart (for progressive disease [PD], 1 to 3 weeks apart). The ordering of the responses was: complete response (CR), partial response (PR), minimal response (MR), no change (NC) and PD. CR was the best response and the poorest response was PD.
Time Frame: every 28 days during treatment period for up to 6 to 8 cycles
Population: Subjects in the ITT population (all subjects who received at least one dose of study drug and who had at least one post baseline efficacy parameter) were included.
Measure: Number; unit: participants
Arm/Group | VAD Treatment | PAD Treatment
Number analyzed (Participants) | 15 | 13
participants
  CR | 0 | 1
  PR | 5 | 6
  Response Rate (CR + PR) | 5 | 7
  MR | 2 | 0
  Overall Response (CR + PR + MR) | 7 | 7
  NC | 3 | 1
  PD | 1 | 1
  Unknown/Unable to Assess | 4 | 4

2. Primary Outcome: Best Reported Disease Response
Description: The primary efficacy analysis was based on the best response obtained during the treatment period according to the EBMT criteria as assessed by the investigator. The ordering of the responses was: CR, PR, MR, NC and PD. CR was the best response and the poorest response was PD.
Time Frame: every 28 days during treatment period for up to 6 to 8 cycles
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | VAD Treatment | PAD Treatment
Number analyzed (Participants) | 15 | 13
participants
  CR | 1 | 3
  PR | 6 | 4
  Response Rate (CR + PR) | 7 | 7
  MR | 2 | 3
  Overall Response (CR + PR + MR) | 9 | 10
  NC | 5 | 3
  PD | 0 | 0
  Unknown/Unable to Assess | 1 | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the duration from the date of the best confirmed response for subjects who achieved CR or PR to the date of first documented evidence of PD (or relapse for subjects who experienced CR) over the duration of the study. DOR = ([Date of PD or date of censoring - Date of best response]+1)/30.44.
Time Frame: every 28 days during treatment period for up to 6 to 8 cycles
Population: Subjects in the ITT population (all subjects who received at least one dose of study drug and who had at least one post baseline efficacy parameter) were included.There was insufficient data to perform Kaplan Meier analysis (data available for 5 subjects in the VAD group and 6 subjects in the PAD group).
Measure: Number; unit: months
Arm/Group | VAD Treatment | PAD Treatment
Number analyzed (Participants) | 5 | 6
months
  patient 1 | 1.68 [1.68 to 6.18] | 2.83 [2.83 to 7.69]
  patient 2 | 6.18 | 7.69
  patient 3 | 3.71 | 5.52
  patient 4 | 5.42 | 6.57
  patient 5 | 4.73 | 4.96
  patient 6 | NA — only 5 patients have been analyzed in this arm | 7.42

ADVERSE EVENTS:
Time Frame: For up to 6 to 8 cycles, consisting of 28 days each, and for up to a 1-year follow-up period
Arm/Group | VAD Treatment | PAD Treatment
Serious Adverse Events (participants affected / at risk) | 6/16 | 5/13
Other Adverse Events (participants affected / at risk) | 15/16 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAD Treatment (N=16) | PAD Treatment (N=13)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAD Treatment (N=16) | PAD Treatment (N=13)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bronchitis acute (Infections and infestations) | 2 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (4) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 2 (2)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 4 (11) | 2 (7)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (9) | 1 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 2 (4)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (4)
Thrombophlebitis (Vascular disorders) | 1 (2) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to a substantial decline in the use of the VAD regimen as standard of care, recruitment of the study was halted at 30 subjects. It was not possible to statistically evaluate any long term efficacy parameter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days